CLINICAL TRIAL: NCT06190496
Title: Role of Cervical Volume and 3 D Power Doppler Indices for Prediction of Preterm Labour
Brief Title: Cervical Volume and Prediction of Preterm Labor
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Mohamed Galal, Doctor, Assiut University
Other Study IDs: Cervical volume preterm labor
Record Dates: First submitted 2023-12-18; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Preterm Labor; Cervical Volume
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of this research is to assess the predictive value of 3D cervical volume and 3D power Doppler indices in predicting pregnancies at risk of preterm labor.

Secondary aim: to compare 2D cervical length and 3D cervical length in coronal view for predicting preterm labour.

ELIGIBILITY:
Inclusion Criteria:

1. Age : 18-35 years old
2. Singleton pregnancy
3. Gestational age : 18-26 Ws knowing last menstrual period and history of regular mense.

Exclusion Criteria:

1. Multiple gestations (e.g., twins, triplets).
2. History of cervical surgery or cervical cerclage.
3. Known uterine anomalies that could affect cervical assessment.
4. Contraindications for transvaginal ultrasound, such as active vaginal bleeding or infection.
5. Severe fetal anomalies or conditions incompatible with life

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: Pregnant women in the second trimester knowing last menstrual period and history of regular menses at Women's Health Hospital Assuit University
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-20 (Estimated); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
The primary outcome could be the incidence of preterm birth (i.e., births occurring before 37 weeks of gestation) among the study participants. | Baseline
  Obstetric ultrasound:Trans abdominal and trans vaginal ultrasounds will be performed to all of ladies. During the trans vaginal scan, The Pulsatility Index (PI) of the uterine artery and the cervical length will be measured. All ultrasound exams will be performed by a single investigator utilizing GE (voluson S 8) ultrasonography machines with pulsed and color Doppler capabilities (GE Medical Systems, Zipf, Austria).
  Cervical length measurements: The distance between the internal and external os will be measured. For the purposes of this study, at least two CL measurements were performed, with the shorter of the two being used in the analysis.
  Uterine artery Doppler:. The left and right uterine arteries will be measured using trans vaginal ultrasonography with color flow imaging

SECONDARY OUTCOMES:
1. Gestational Age at Delivery: Measure the gestational age at which participants in the study give birth. This information can help assess whether ultrasonic assessments correlate with the timing of delivery. | Baseline
  Obstetric ultrasound:Trans abdominal and trans vaginal ultrasounds will be performed to all of ladies. During the trans vaginal scan, The Pulsatility Index (PI) of the uterine artery and the cervical length will be measured. All ultrasound exams will be performed by a single investigator utilizing GE (voluson S 8) ultrasonography machines with pulsed and color Doppler capabilities (GE Medical Systems, Zipf, Austria).
  Cervical length measurements: The distance between the internal and external os will be measured. For the purposes of this study, at least two CL measurements were performed, with the shorter of the two being used in the analysis.
  Uterine artery Doppler:. The left and right uterine arteries will be measured using trans vaginal ultrasonography with color flow imaging
2. Predictive Parameters: Analyse the individual and combined predictive power of cervical length, vascularity indices, and cervical volume. Determine which of these parameters (or their combinations) show the strongest correlation with preterm birth | Baseline
  Obstetric ultrasound:Trans abdominal and trans vaginal ultrasounds will be performed to all of ladies. During the trans vaginal scan, The Pulsatility Index (PI) of the uterine artery and the cervical length will be measured. All ultrasound exams will be performed by a single investigator utilizing GE (voluson S 8) ultrasonography machines with pulsed and color Doppler capabilities (GE Medical Systems, Zipf, Austria).
  Cervical length measurements: The distance between the internal and external os will be measured. For the purposes of this study, at least two CL measurements were performed, with the shorter of the two being used in the analysis.
  Uterine artery Doppler:. The left and right uterine arteries will be measured using trans vaginal ultrasonography with color flow imaging